CLINICAL TRIAL: NCT05297630
Title: Comparative Evaluation of the Evolution of Emerging Biological Markers (sST2, Copeptin, Chromogranin, NGAL, suPAR and Cystatin) in Patients Hospitalized for Acute Heart Failure (AHF) Depending on Their Management: Conventional or Therapeutic Adjustment According to Daily Ultrasound. Ancillary Study to the JECICA Study (AOI GCS MERRI 2015).
Brief Title: Comparative Evaluation of the Evolution of Emerging Biological Markers in Patients Hospitalized for Acute Heart Failure According to Conventional Management or Therapeutic Adjustment Via Daily Ultrasound.
Acronym: JECICA2
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: AOI/2020/JET01
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Heart Failure
Keywords: Heart failure; hospitalization; biomarkers; sST2; prognosis; therapeutic
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The samples analyzed in the JECICA2 study come from the serum library already constituted from the population of the original JECICA study, the selection criteria of which are as follows (samples available from 169 patients, collected at D0 and 1 month).
  Patients hospitalized for acute heart failure who received at least 40mg of IV furosemide.
  Patients with impaired Left Ventricular Ejection Fraction, <50%. Patients with an Nt-ProBNP value >1200pg/ml.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Jet Echo group: Biological markers from heart failure patients who underwent therapeutic adjustment according to a daily ultrasound scan
  Interventions: Other: Evaluation of the evolution of biological markers from the biobank.
- Conventional management group: Biological markers from heart failure patients who had conventional management.
  Interventions: Other: Evaluation of the evolution of biological markers from the biobank.

INTERVENTIONS:
Other: Evaluation of the evolution of biological markers from the biobank. — The evolution of sST2, copeptin, chromogranin, NGAL, suPAR and cystatin will be evaluated between Day 0 and Month 1

SUMMARY:
This is a bi-centric, prospective randomized study to evaluate the contribution of rapid echocardioscopy at the patient's bedside to improving the prognosis of patients hospitalized for acute heart failure. The following markers will be evaluated: sST2, Copeptin, chromogranin, NGAL, suPAR and cystatin.

DETAILED DESCRIPTION:
The JECICA study is the first prospective randomized study to evaluate the contribution of rapid echocardioscopy at the patient's bedside to improving the prognosis of patients hospitalized for acute heart failure (paper submitted to the American Heart Journal, Impact Factor 4.15). The serum library set up to consider this ancillary study can now be used.

With it, a comparative analysis of the expression profiles of emerging biological markers will be made according to whether patients received standard management or the "Jet Echo" strategy. The following markers will be evaluated: sST2, Copeptin, chromogranin, NGAL, suPAR and cystatin. This study should help to explain any differences in results observed, consider the development of multiparametric prognostic scores and explore the correlation between biological markers and the evaluation of echocardiographic congestion from a pathophysiological viewpoint.

The results obtained should lead us to improve our usual practices for the management of heart failure patients.

ELIGIBILITY:
Inclusion Criteria: (General inclusion criteria)

* The patient or his representative must have given free and informed consent and signed the consent form.
* The patient must be affiliated to or beneficiary of a health insurance plan.
* The patient must have been available for 6 months of follow-up.
* The patient is at least (>) 18 years of age.

Inclusion criteria for target population:

* Patient hospitalized for acute heart failure who received at least 40mg of IV furosemide.
* Patient with impaired Left Ventricle Ejection Fraction <50%.
* Patient with an Nt-ProBNP value >1200pg/ml.

Exclusion Criteria : (General non-inclusion criteria)

* Subject is participating in another study.
* Subject is in an exclusion period determined by a previous study.
* Subject is under court protection.
* Subject or subject's representative refuses to sign consent.
* It is not possible to provide the subject or the subject's representative with informed information.

Criteria for non-inclusion regarding associated interfering diseases or conditions:

* Patient is pregnant or breastfeeding.
* Patient is already included in a surveillance program (PRADO, OSICAT).
* Patient has a mechanical or biological mitral prosthesis.
* History of mitral narrowing.
* Severe valve disease with a surgical deadline within a month (<30 days).
* Chronic renal failure on dialysis.
* High grade BAV (BAV 2/1 and BAV3).
* Hypertrophic cardiomyopathy.
* Cardiogenic shock.
* Contraindication to furosemide.
* Anechoic patient.

Exclusion criteria:

- Patient hospitalized for more than (>) 1 month.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Serum library already constituted from the population of the original JECICA study whose selection criteria are described above (samples available from 169 patients, collected at D0 and at 1 month).
Sampling Method: Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-07-09 (Actual); Study Completion 2022-07-09 (Actual)

PRIMARY OUTCOMES:
Evolution of the emerging biological marker sST2 in plasma samples from the Jet Echo group. | Day 0
  Quantitative, ng/mL
Evolution of the emerging biological marker sST2 in plasma samples from the Jet Echo group. | 1 Month
  Quantitative, ng/mL
Evolution of the emerging biological marker sST2 in plasma samples from the conventional management group. | Day 0
  Quantitative, ng/mL
Evolution of the emerging biological marker sST2 in plasma samples from the conventional management group. | 1 Month
  Quantitative, ng/mL
Evolution of the emerging biological marker copeptin in plasma samples from the Jet Echo group | Day 0
  Quantitative, pmol/L
Evolution of the emerging biological marker copeptin in plasma samples from the Jet Echo group | Month 1
  Quantitative, pmol/L
Evolution of the emerging biological marker copeptin in plasma samples from the conventional management group | Day 0
  Quantitative, pmol/L
Evolution of the emerging biological marker copeptin in plasma samples from the conventional management group | Month 1
  Quantitative, pmol/L
Evolution of the emerging biological marker chromogranin in plasma samples from the Jet Echo group | Day 0
  Quantitative, ng/mL
Evolution of the emerging biological marker chromogranin in plasma samples from the Jet Echo group | Month 1
  Quantitative, ng/mL
Evolution of the emerging biological marker chromogranin in plasma samples from the conventional management group | Day 0
  Quantitative, ng/mL
Evolution of the emerging biological marker chromogranin in plasma samples from the conventional management group | Month 1
  Quantitative, ng/mL
Evolution of the emerging biological marker NGAL in plasma samples from the Jet Echo group. | Day 0
  Quantitative, ng/mL
Evolution of the emerging biological marker NGAL in plasma samples from the Jet Echo group. | Month 1
  Quantitative, ng/mL
Evolution of the emerging biological marker NGAL in plasma samples from the conventional management group. | Day 0
  Quantitative, ng/mL
Evolution of the emerging biological marker NGAL in plasma samples from the conventional management group. | Month 1
  Quantitative, ng/mL
Evolution of the emerging biological marker suPAR in plasma samples from the Jet Echo group. | Day 0
  Quantitative, ng/mL
Evolution of the emerging biological marker suPAR in plasma samples from the Jet Echo group. | Month 1
  Quantitative, ng/mL
Evolution of the emerging biological marker suPAR in plasma samples from the conventional management group. | Day 0
  Quantitative, ng/mL
Evolution of the emerging biological marker suPAR in plasma samples from the conventional management group. | Month 1
  Quantitative, ng/mL
Evolution of the emerging biological marker cystatin in plasma samples from the Jet Echo group. | Day 0
  Quantitative, ng/mL
Evolution of the emerging biological marker cystatin in plasma samples from the Jet Echo group. | Month 1
  Quantitative, ng/mL
Evolution of the emerging biological marker cystatin in plasma samples from the conventional management group. | Day 0
  Quantitative, ng/mL
Evolution of the emerging biological marker cystatin in plasma samples from the conventional management group. | Month 1
  Quantitative, ng/mL

SECONDARY OUTCOMES:
Correlation between emerging biomarkers and clinical symptomatology in the Jet Echo group: Sex | Day 0
  The sex of participants will be noted as Male/Female
Correlation between emerging biomarkers and clinical symptomatology in the conventional management group: Sex | Day 0
  The sex of participants will be noted as Male/Female
Correlation between emerging biomarkers and clinical symptomatology in the Jet Echo group: Age | Day 0
  The age of participants will be noted in years
Correlation between emerging biomarkers and clinical symptomatology in the conventional management group: Age | Day 0
  The age of participants will be noted in years
Correlation between emerging biomarkers and clinical symptomatology in the Jet Echo group: Diuresis | Day 0
  The diuresis of participants will be measured in millilitres
Correlation between emerging biomarkers and clinical symptomatology in the Jet Echo group: Diuresis | Month 1
  The diuresis of participants will be measured in millilitres
Correlation between emerging biomarkers and clinical symptomatology in the conventional management group: Diuresis | Day 0
  The diuresis of participants will be measured in millilitres
Correlation between emerging biomarkers and clinical symptomatology in the conventional management group: Diuresis | Month 1
  The diuresis of participants will be measured in millilitres
Correlation between emerging biomarkers and clinical symptomatology in the Jet Echo group: blood pressure | Day 0
  The blood pressure of participants will be noted
Correlation between emerging biomarkers and clinical symptomatology in the Jet Echo group: blood pressure | Month 1
  The blood pressure of participants will be noted
Correlation between emerging biomarkers and clinical symptomatology in the conventional management group: blood pressure | Day 0
  The blood pressure of participants will be noted
Correlation between emerging biomarkers and clinical symptomatology in the conventional management group: blood pressure | Month 1
  The blood pressure of participants will be noted
Correlation between emerging biomarkers and clinical symptomatology in the Jet Echo group: heart rate | Day 0
  The heart rate of participants will be noted
Correlation between emerging biomarkers and clinical symptomatology in the Jet Echo group: heart rate | Month 1
  The heart rate of participants will be noted
Correlation between emerging biomarkers and clinical symptomatology in the conventional management group: heart rate | Day 0
  The heart rate of participants will be noted
Correlation between emerging biomarkers and clinical symptomatology in the conventional management group: heart rate | Month 1
  The heart rate of participants will be noted
Correlation between emerging biomarkers and clinical symptomatology in the Jet Echo group: risk factors | Day 0
  Cardiovascular risk factors (hypertension, diabetes, dyslipidemia, heredity) will be noted
Correlation between emerging biomarkers and clinical symptomatology in the Jet Echo group: risk factors | Month 1
  Cardiovascular risk factors (hypertension, diabetes, dyslipidemia, heredity) will be noted
Correlation between emerging biomarkers and clinical symptomatology in the conventional management group: risk factors | Day 0
  Cardiovascular risk factors (hypertension, diabetes, dyslipidemia, heredity) will be noted
Correlation between emerging biomarkers and clinical symptomatology in the conventional management group: risk factors | Month 1
  Cardiovascular risk factors (hypertension, diabetes, dyslipidemia, heredity) will be noted
Correlation between emerging biomarkers and clinical symptomatology in the Jet Echo group: history | Day 0
  The history and etiology of the heart disease (ischemic dilated, rhythmic, valvular, toxic, alcoholic) will be noted.
Correlation between emerging biomarkers and clinical symptomatology in the Jet Echo group: history | Month 1
  The history and etiology of the heart disease (ischemic dilated, rhythmic, valvular, toxic, alcoholic) will be noted.
Correlation between emerging biomarkers and clinical symptomatology in the conventional management group: history | Day 0
  The history and etiology of the heart disease (ischemic dilated, rhythmic, valvular, toxic, alcoholic) will be noted.
Correlation between emerging biomarkers and clinical symptomatology in the conventional management group: history | Month 1
  The history and etiology of the heart disease (ischemic dilated, rhythmic, valvular, toxic, alcoholic) will be noted.
Correlation between emerging biomarkers and clinical symptomatology in the Jet Echo group: Left ventricle Ejection Fraction | Day 0
  The Left ventricle Ejection Fraction will be measured as a %.
Correlation between emerging biomarkers and clinical symptomatology in the Jet Echo group: Left ventricle Ejection Fraction | Month 1
  The Left ventricle Ejection Fraction will be measured as a %.
Correlation between emerging biomarkers and clinical symptomatology in the conventional management group: Left ventricle Ejection Fraction | Day 0
  The Left ventricle Ejection Fraction will be measured as a %.
Correlation between emerging biomarkers and clinical symptomatology in the conventional management group: Left ventricle Ejection Fraction | Month 1
  The Left ventricle Ejection Fraction will be measured as a %.
Correlation between emerging biomarkers and clinical symptomatology in the Jet Echo group: renal insufficiency stage | Day 0
  The stage of renal insufficiency (urea, creatinine, Calcium-Dependent Protein Kinase clearance) will be measured.
Correlation between emerging biomarkers and clinical symptomatology in the Jet Echo group: renal insufficiency stage | Month 1
  The stage of renal insufficiency (urea, creatinine, Calcium-Dependent Protein Kinase clearance) will be measured.
Correlation between emerging biomarkers and clinical symptomatology in the conventional management group: renal insufficiency stage | Day 0
  The stage of renal insufficiency (urea, creatinine, Calcium-Dependent Protein Kinase clearance) will be measured.
Correlation between emerging biomarkers and clinical symptomatology in the conventional management group: renal insufficiency stage | Month 1
  The stage of renal insufficiency (urea, creatinine, Calcium-Dependent Protein Kinase clearance) will be measured.
Correlation between emerging biomarkers and clinical symptomatology in the Jet Echo group: New York Heart Association stage | Day 0
  The New York Heart Association stage will be noted
Correlation between emerging biomarkers and clinical symptomatology in the Jet Echo group: New York Heart Association stage | Month 1
  The New York Heart Association stage will be noted
Correlation between emerging biomarkers and clinical symptomatology in the conventional management group: New York Heart Association stage | Day 0
  The New York Heart Association stage will be noted
Correlation between emerging biomarkers and clinical symptomatology in the conventional management group: New York Heart Association stage | Month 1
  The New York Heart Association stage will be noted
Correlation between emerging biomarkers and clinical symptomatology in the Jet Echo group: Type of heart failure | Day 0
  The type of heart failure (congestive heart failure/left heart failure/right heart failure) will be noted
Correlation between emerging biomarkers and clinical symptomatology in the Jet Echo group: Type of heart failure | Month 1
  The type of heart failure (congestive heart failure/left heart failure/right heart failure) will be noted
Correlation between emerging biomarkers and clinical symptomatology in the conventional management group: Type of heart failure | Day 0
  The type of heart failure (congestive heart failure/left heart failure/right heart failure) will be noted
Correlation between emerging biomarkers and clinical symptomatology in the conventional management group: Type of heart failure | Month 1
  The type of heart failure (congestive heart failure/left heart failure/right heart failure) will be noted
Correlation between emerging biomarkers and clinical symptomatology in the Jet Echo group: Type of therapy | Day 0
  The therapy given (Beta-blocker, ACE inhibitor, ARB2, Anti aldosterone, diuretics) and dosage, Implantable cardiac device, pacemaker will be noted.
Correlation between emerging biomarkers and clinical symptomatology in the Jet Echo group: Type of therapy | Month 1
  The therapy given (Beta-blocker, ACE inhibitor, ARB2, Anti aldosterone, diuretics) and dosage, Implantable cardiac device, pacemaker will be noted.
Correlation between emerging biomarkers and clinical symptomatology in the conventional management group: Type of therapy | Day 0
  The therapy given (Beta-blocker, ACE inhibitor, ARB2, Anti aldosterone, diuretics) and dosage, Implantable cardiac device, pacemaker will be noted.
Correlation between emerging biomarkers and clinical symptomatology in the conventional management group: Type of therapy | Month 1
  The therapy given (Beta-blocker, ACE inhibitor, ARB2, Anti aldosterone, diuretics) and dosage, Implantable cardiac device, pacemaker will be noted.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Nîmes University Hospital, Nîmes, Gard
  - Montpellier University Hospital, Arnaud de Villeneuve, Montpellier, Hérault

REFERENCES:
- [Background] Brennan JM, Blair JE, Goonewardena S, Ronan A, Shah D, Vasaiwala S, Brooks E, Levy A, Kirkpatrick JN, Spencer KT. A comparison by medicine residents of physical examination versus hand-carried ultrasound for estimation of right atrial pressure. Am J Cardiol. 2007 Jun 1;99(11):1614-6. doi: 10.1016/j.amjcard.2007.01.037. Epub 2007 Apr 18. PMID 17531592
- [Background] Capomolla S, Ceresa M, Pinna G, Maestri R, La Rovere MT, Febo O, Rossi A, Paganini V, Caporotondi A, Guazzotti G, Gnemmi M, Mortara A, Cobelli F. Echo-Doppler and clinical evaluations to define hemodynamic profile in patients with chronic heart failure: accuracy and influence on therapeutic management. Eur J Heart Fail. 2005 Jun;7(4):624-30. doi: 10.1016/j.ejheart.2004.07.013. PMID 15921804
- [Background] Chakko S, Woska D, Martinez H, de Marchena E, Futterman L, Kessler KM, Myerberg RJ. Clinical, radiographic, and hemodynamic correlations in chronic congestive heart failure: conflicting results may lead to inappropriate care. Am J Med. 1991 Mar;90(3):353-9. doi: 10.1016/0002-9343(91)80016-f. PMID 1825901
- [Background] Gheorghiade M, Pang PS. Acute heart failure syndromes. J Am Coll Cardiol. 2009 Feb 17;53(7):557-573. doi: 10.1016/j.jacc.2008.10.041. PMID 19215829
- [Background] Go AS, Mozaffarian D, Roger VL, Benjamin EJ, Berry JD, Blaha MJ, Dai S, Ford ES, Fox CS, Franco S, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Huffman MD, Judd SE, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Mackey RH, Magid DJ, Marcus GM, Marelli A, Matchar DB, McGuire DK, Mohler ER 3rd, Moy CS, Mussolino ME, Neumar RW, Nichol G, Pandey DK, Paynter NP, Reeves MJ, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Executive summary: heart disease and stroke statistics--2014 update: a report from the American Heart Association. Circulation. 2014 Jan 21;129(3):399-410. doi: 10.1161/01.cir.0000442015.53336.12. No abstract available. PMID 24446411
- [Background] Goonewardena SN, Spencer KT. Handcarried echocardiography to assess hemodynamics in acute decompensated heart failure. Curr Heart Fail Rep. 2010 Dec;7(4):219-27. doi: 10.1007/s11897-010-0030-8. PMID 20890689
- [Background] Heidenreich PA, Trogdon JG, Khavjou OA, Butler J, Dracup K, Ezekowitz MD, Finkelstein EA, Hong Y, Johnston SC, Khera A, Lloyd-Jones DM, Nelson SA, Nichol G, Orenstein D, Wilson PW, Woo YJ; American Heart Association Advocacy Coordinating Committee; Stroke Council; Council on Cardiovascular Radiology and Intervention; Council on Clinical Cardiology; Council on Epidemiology and Prevention; Council on Arteriosclerosis; Thrombosis and Vascular Biology; Council on Cardiopulmonary; Critical Care; Perioperative and Resuscitation; Council on Cardiovascular Nursing; Council on the Kidney in Cardiovascular Disease; Council on Cardiovascular Surgery and Anesthesia, and Interdisciplinary Council on Quality of Care and Outcomes Research. Forecasting the future of cardiovascular disease in the United States: a policy statement from the American Heart Association. Circulation. 2011 Mar 1;123(8):933-44. doi: 10.1161/CIR.0b013e31820a55f5. Epub 2011 Jan 24. PMID 21262990
- [Background] Huet F, Nicoleau J, Dupuy AM, Curinier C, Breuker C, Castet-Nicolas A, Lotierzo M, Kalmanovich E, Zerkowski L, Akodad M, Adda J, Agullo A, Leclercq F, Pasquie JL, Battistella P, Roubille C, Fesler P, Mercier G, Bourel G, Cristol JP, Roubille F. STADE-HF (sST2 As a help for management of HF): a pilot study. ESC Heart Fail. 2020 Apr;7(2):774-778. doi: 10.1002/ehf2.12663. Epub 2020 Mar 13. PMID 32168423
- [Background] Lei J, Dhamoon AS, Wang J, Iannuzzi M, Liu K. Walking the tightrope: Using quantitative Doppler echocardiography to optimize ventricular filling pressures in patients hospitalized for acute heart failure. Eur Heart J Acute Cardiovasc Care. 2016 Apr;5(2):130-40. doi: 10.1177/2048872615573517. Epub 2015 Feb 18. PMID 25694508
- [Background] Lotierzo M, Dupuy AM, Kalmanovich E, Roubille F, Cristol JP. sST2 as a value-added biomarker in heart failure. Clin Chim Acta. 2020 Feb;501:120-130. doi: 10.1016/j.cca.2019.10.029. Epub 2019 Oct 31. PMID 31678574
- [Background] McMurray JJ, Adamopoulos S, Anker SD, Auricchio A, Bohm M, Dickstein K, Falk V, Filippatos G, Fonseca C, Gomez-Sanchez MA, Jaarsma T, Kober L, Lip GY, Maggioni AP, Parkhomenko A, Pieske BM, Popescu BA, Ronnevik PK, Rutten FH, Schwitter J, Seferovic P, Stepinska J, Trindade PT, Voors AA, Zannad F, Zeiher A; Task Force for the Diagnosis and Treatment of Acute and Chronic Heart Failure 2012 of the European Society of Cardiology; Bax JJ, Baumgartner H, Ceconi C, Dean V, Deaton C, Fagard R, Funck-Brentano C, Hasdai D, Hoes A, Kirchhof P, Knuuti J, Kolh P, McDonagh T, Moulin C, Popescu BA, Reiner Z, Sechtem U, Sirnes PA, Tendera M, Torbicki A, Vahanian A, Windecker S, McDonagh T, Sechtem U, Bonet LA, Avraamides P, Ben Lamin HA, Brignole M, Coca A, Cowburn P, Dargie H, Elliott P, Flachskampf FA, Guida GF, Hardman S, Iung B, Merkely B, Mueller C, Nanas JN, Nielsen OW, Orn S, Parissis JT, Ponikowski P; ESC Committee for Practice Guidelines. ESC guidelines for the diagnosis and treatment of acute and chronic heart failure 2012: The Task Force for the Diagnosis and Treatment of Acute and Chronic Heart Failure 2012 of the European Society of Cardiology. Developed in collaboration with the Heart Failure Association (HFA) of the ESC. Eur J Heart Fail. 2012 Aug;14(8):803-69. doi: 10.1093/eurjhf/hfs105. No abstract available. PMID 22828712
- [Background] Metra M, Cotter G, Gheorghiade M, Dei Cas L, Voors AA. The role of the kidney in heart failure. Eur Heart J. 2012 Sep;33(17):2135-42. doi: 10.1093/eurheartj/ehs205. Epub 2012 Aug 10. PMID 22888113
- [Background] Nguyen VT, Ho JE, Ho CY, Givertz MM, Stevenson LW. Handheld echocardiography offers rapid assessment of clinical volume status. Am Heart J. 2008 Sep;156(3):537-42. doi: 10.1016/j.ahj.2008.04.015. Epub 2008 Jun 17. PMID 18760138
- [Background] Ovbiagele B, Goldstein LB, Higashida RT, Howard VJ, Johnston SC, Khavjou OA, Lackland DT, Lichtman JH, Mohl S, Sacco RL, Saver JL, Trogdon JG; American Heart Association Advocacy Coordinating Committee and Stroke Council. Forecasting the future of stroke in the United States: a policy statement from the American Heart Association and American Stroke Association. Stroke. 2013 Aug;44(8):2361-75. doi: 10.1161/STR.0b013e31829734f2. Epub 2013 May 22. PMID 23697546
- [Background] Parrinello G, Torres D, Paterna S, Di Pasquale P, Mezzero M, Licata G. The challenge of the volume status assessment in heart failure. Am Heart J. 2009 Apr;157(4):e19-20; author reply e21. doi: 10.1016/j.ahj.2008.12.001. Epub 2009 Jan 31. No abstract available. PMID 19332179
- [Background] Remes J, Miettinen H, Reunanen A, Pyorala K. Validity of clinical diagnosis of heart failure in primary health care. Eur Heart J. 1991 Mar;12(3):315-21. doi: 10.1093/oxfordjournals.eurheartj.a059896. PMID 2040313
- [Background] Ricci JE, Kalmanovich E, Robert C, Chevallier T, Aguilhon S, Solecki K, Akodad M, Cornillet L, Soullier C, Cayla G, Lattuca B, Roubille F. Management of acute heart failure: Contribution of daily bedside echocardiographic assessment on therapy adjustment with impact measure on the 30-day readmission rate (JECICA). Contemp Clin Trials Commun. 2018 Aug 9;12:103-108. doi: 10.1016/j.conctc.2018.07.006. eCollection 2018 Dec. PMID 30364633
- [Background] Ronco C, Cicoira M, McCullough PA. Cardiorenal syndrome type 1: pathophysiological crosstalk leading to combined heart and kidney dysfunction in the setting of acutely decompensated heart failure. J Am Coll Cardiol. 2012 Sep 18;60(12):1031-42. doi: 10.1016/j.jacc.2012.01.077. Epub 2012 Jul 25. PMID 22840531
- [Background] Ross JS, Chen J, Lin Z, Bueno H, Curtis JP, Keenan PS, Normand SL, Schreiner G, Spertus JA, Vidan MT, Wang Y, Wang Y, Krumholz HM. Recent national trends in readmission rates after heart failure hospitalization. Circ Heart Fail. 2010 Jan;3(1):97-103. doi: 10.1161/CIRCHEARTFAILURE.109.885210. Epub 2009 Nov 10. PMID 19903931
- [Background] Stewart S, MacIntyre K, Hole DJ, Capewell S, McMurray JJ. More 'malignant' than cancer? Five-year survival following a first admission for heart failure. Eur J Heart Fail. 2001 Jun;3(3):315-22. doi: 10.1016/s1388-9842(00)00141-0. PMID 11378002
- [Background] Tuppin P, Cuerq A, de Peretti C, Fagot-Campagna A, Danchin N, Juilliere Y, Alla F, Allemand H, Bauters C, Drici MD, Hagege A, Jondeau G, Jourdain P, Leizorovicz A, Paccaud F. Two-year outcome of patients after a first hospitalization for heart failure: A national observational study. Arch Cardiovasc Dis. 2014 Mar;107(3):158-68. doi: 10.1016/j.acvd.2014.01.012. Epub 2014 Mar 21. PMID 24662470
- [Background] Vitarelli A, Gheorghiade M. Transthoracic and transesophageal echocardiography in the hemodynamic assessment of patients with congestive heart failure. Am J Cardiol. 2000 Aug 17;86(4A):36G-40G. doi: 10.1016/s0002-9149(00)00990-5. PMID 10997352
- [Background] Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Drazner MH, Fonarow GC, Geraci SA, Horwich T, Januzzi JL, Johnson MR, Kasper EK, Levy WC, Masoudi FA, McBride PE, McMurray JJ, Mitchell JE, Peterson PN, Riegel B, Sam F, Stevenson LW, Tang WH, Tsai EJ, Wilkoff BL; American College of Cardiology Foundation; American Heart Association Task Force on Practice Guidelines. 2013 ACCF/AHA guideline for the management of heart failure: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2013 Oct 15;62(16):e147-239. doi: 10.1016/j.jacc.2013.05.019. Epub 2013 Jun 5. No abstract available. PMID 23747642